CLINICAL TRIAL: NCT00005318
Title: ARDS - Clinical Epidemiology and the Role of the Inflammatory Response - SCOR in Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4091; P50HL050152 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Diseases
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases

SUMMARY:
To investigate the epidemiology of adult respiratory distress syndrome (ARDS) and the evolution of the inflammatory process in patients with acute lung injury.

DETAILED DESCRIPTION:
BACKGROUND:

The results provided: a) a better understanding of the evolution of inflammation in clinical conditions leading to lung injury; b) a better understanding of the mechanisms of the initial injury and its propagation; and c) information that will help predict the course and outcome in individual patients. These data should be useful in guiding the choice and timing of specific therapeutic interventions.

DESIGN NARRATIVE:

The study was a subproject within a Specialized Center of Research (SCOR) in Acute Lung Injury. Leonard Hudson was the subproject principal investigator. The epidemiological aspects focussed on refining clinical criteria that predicted patients at high risk for the onset of ARDS, and identifying these patients as early as possible before the onset of lung injury. The major hypothesis was that uncontrolled and sustained alveolar inflammation increased the severity of ARDS and prolonged its course, and that sustained inflammation was more likely to occur when ARDS followed sepsis syndrome than multiple trauma. The investigators also tested the hypothesis that the pattern of the inflammatory response in blood and lungs was an important determinant of whether lung inflammation persisted or resolved. Important components of the inflammatory response studied included; 1) a coordinated sequence of cytokines in blood and lung lavage fluid; 2) the expression of adhesion molecules on blood leukocytes; 3) circulating markers of diffuse endothelial injury (VWF and ELAM1); 4) products of the arachidonic acid cascade; 5) the induction of endogenous proteins that modified the host response to bacterial products such as endotoxin; and 6) inflammatory cell populations and proteins in the lung. Patterns of inflammation were correlated with clinical risks, critical clinical events, and outcome measures.

The study was renewed in 1999 to : develop clinical prediction tools that provide individual risk assessment for the onset and outcome of lung injury; determine the incidence and outcome of acute lung injury / adult respiratory distress syndrome (ALI/ARDS) in populations beyond a single institution; determine the relationship between inflammatory responses and injury to the lung endothelial and epithelial barriers; and investigate determinants of host susceptibility that modulate the occurrence of ALI/ARDS in patients at risk.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-01; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Hudson — University of Washington

REFERENCES:
- [Background] Hudson LD, Milberg JA, Anardi D, Maunder RJ. Clinical risks for development of the acute respiratory distress syndrome. Am J Respir Crit Care Med. 1995 Feb;151(2 Pt 1):293-301. doi: 10.1164/ajrccm.151.2.7842182.
- [Background] Davidson TA, Rubenfeld GD, Caldwell ES, Hudson LD, Steinberg KP. The effect of acute respiratory distress syndrome on long-term survival. Am J Respir Crit Care Med. 1999 Dec;160(6):1838-42. doi: 10.1164/ajrccm.160.6.9903058. PMID 10588594
- [Background] Davidson TA, Caldwell ES, Curtis JR, Hudson LD, Steinberg KP. Reduced quality of life in survivors of acute respiratory distress syndrome compared with critically ill control patients. JAMA. 1999 Jan 27;281(4):354-60. doi: 10.1001/jama.281.4.354. PMID 9929089
- [Background] Madtes DK, Rubenfeld G, Klima LD, Milberg JA, Steinberg KP, Martin TR, Raghu G, Hudson LD, Clark JG. Elevated transforming growth factor-alpha levels in bronchoalveolar lavage fluid of patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 1998 Aug;158(2):424-30. doi: 10.1164/ajrccm.158.2.9711112. PMID 9700116
- [Background] Matute-Bello G, Liles WC, Radella F 2nd, Steinberg KP, Ruzinski JT, Jonas M, Chi EY, Hudson LD, Martin TR. Neutrophil apoptosis in the acute respiratory distress syndrome. Am J Respir Crit Care Med. 1997 Dec;156(6):1969-77. doi: 10.1164/ajrccm.156.6.96-12081. PMID 9412582
- [Background] Kurdowska A, Noble JM, Steinberg KP, Ruzinski J, Hudson LD, Martin TR. Anti-IL-8 autoantibodies in alveolar fluid from patients at risk for ARDS and with well-defined ARDS. Chest. 1999 Jul;116(1 Suppl):9S. doi: 10.1378/chest.116.suppl_1.9s. No abstract available. PMID 10424560
- [Background] Moss M, Parsons PE, Steinberg KP, Hudson LD, Guidot DM, Burnham EL, Eaton S, Cotsonis GA. Chronic alcohol abuse is associated with an increased incidence of acute respiratory distress syndrome and severity of multiple organ dysfunction in patients with septic shock. Crit Care Med. 2003 Mar;31(3):869-77. doi: 10.1097/01.CCM.0000055389.64497.11. PMID 12626999
- [Background] Treggiari MM, Hudson LD, Martin DP, Weiss NS, Caldwell E, Rubenfeld G. Effect of acute lung injury and acute respiratory distress syndrome on outcome in critically ill trauma patients. Crit Care Med. 2004 Feb;32(2):327-31. doi: 10.1097/01.CCM.0000108870.09693.42. PMID 14758144
- [Background] Johnston CJ, Rubenfeld GD, Hudson LD. Effect of age on the development of ARDS in trauma patients. Chest. 2003 Aug;124(2):653-9. doi: 10.1378/chest.124.2.653. PMID 12907556
- [Background] Rubenfeld GD, Cooper C, Carter G, Thompson BT, Hudson LD. Barriers to providing lung-protective ventilation to patients with acute lung injury. Crit Care Med. 2004 Jun;32(6):1289-93. doi: 10.1097/01.ccm.0000127266.39560.96. PMID 15187508